CLINICAL TRIAL: NCT06444984
Title: The Movie Theater Study: Acute Cardiometabolic Effects of a Cinema-Style Meal
Brief Title: The Movie Theater Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2141491-1
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Hyperglycemia, Postprandial; Hyperinsulinemia
MeSH Terms: conditions — Hyperglycemia; Hyperinsulinism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting Meal Trial (Experimental): During the fasting meal trial, participants will report fasted and consume a movie theater style meal.
  Interventions: Other: Fasting Trial
- Fed Meal Trial (Experimental): During the fed meal trial, participants will report fasted and first consume a high-fat breakfast. Participants will then be asked to consume a movie theater style meal three hours later.
  Interventions: Other: Fed Trial

INTERVENTIONS:
Other: Fasting Trial — Participants will report fasted and consume popcorn (6 cups popped microwave popcorn), soda (32 oz Coke-a-cola), and candy (2.17 oz of Skittles) in the morning.
  Arms: Fasting Meal Trial
Other: Fed Trial — Participants will report fasted and first consume a high-fat meal (Jimmy Deans) in the morning. After a three-hour break, participants will consume popcorn (6 cups popped microwave popcorn), soda (32 oz Coke-a-cola), and candy (2.17 oz of Skittles).
  Arms: Fed Meal Trial

SUMMARY:
Increasing attention has been paid to meals with unusual characteristics that are consumed on a semi-regular basis (e.g., "tailgating," pizza buffets). The purpose of this study is to describe the acute cardiometabolic effects of a cinema-style meal rich in refined sugar, total carbohydrate, and moderate in fat (i.e., soda, popcorn, candy).

DETAILED DESCRIPTION:
Participants will complete two study visits in random order. For one visit, participants will consume popcorn (6 cups popped microwave popcorn), soda (32 oz Coke-a-cola), and candy (2.17 oz of Skittles) in the morning while fasting (i.e., the "fasting trial"). For the other visit, participants will report fasting and then first consume a high-fat meal (two Jimmy Dean's breakfast sandwiches; the "fed trial"). After consuming the high-fat meal during the fed trial, participants will be allowed to leave for three hours. During this three-hour period, the investigators will ask participants to only consume water and remain sedentary. Upon return, participants will consume the same movie theater style meal (popcorn, soda, candy).

Regardless of fasting or fed trials, procedures for this study will be largely similar between the two visits. Participants will arrive having fasted for ~10 hours, avoided exercise and alcohol for > 24 hours, and avoided anti-inflammatory medications for > 72 hours. First, the investigators will perform a baseline vascular ultrasound using the flow-mediated dilation (FMD) technique on all participants. Upon completion of FMD, the investigators will perform a blood draw in one of two ways (depending on the trial). For the fasting trial, the investigators will insert an indwelling intravenous catheter (IV) to minimize needle sticks. After a baseline blood sample is collected, participants will consume the movie theater-style meal and remain in the lab for four hours. During this time, the investigators will collect blood samples at 0.5-, 1-, 2-, 3-, and 4-hours post meal to measure potential changes in metabolic and inflammatory markers and indicators of endotoxemia. The investigators will also measure FMD at 2- and 4-hours post movie theater-style meal. During the fed trial, the investigators will first perform a single venipuncture to obtain a blood sample in order to have a true baseline sample for the fed trial. When participants return from this three-hour break, the procedures for the fed trial will be identical to the fasting trial (IV inserted, moving theater meal consumed, serial blood draws and FMD completed at the same timepoints over a four-hour period).

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Not pregnant or expecting to become pregnant (females only)
* Not postmenopausal (females only).
* Not been diagnosed with a cardiometabolic conditions (e.g., heart disease, type 2 diabetes)
* Not been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* Does not regularly take anti-inflammatory drugs (more than 2x week) or able to temporarily suspend use of anti-inflammatory drugs.
* Does not use glucose-lowering drugs (e.g., metformin)
* Does not use lipid-lowering drugs (e.g., statins)
* Does not use tobacco products or any illicit drugs.
* Does not have a pacemaker.

Exclusion Criteria:

* Not 18-45 years old
* Pregnant or expecting to become pregnant (females only)
* Postmenopausal (females only).
* Been diagnosed with a cardiometabolic conditions (e.g., heart disease, type 2 diabetes)
* Been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* Regularly take anti-inflammatory drugs (more than 2x week) or unable to temporarily suspend use of anti-inflammatory drugs.
* Use glucose-lowering drugs (e.g., metformin)
* Use lipid-lowering drugs (e.g., statins)
* Use tobacco products or any illicit drugs.
* Has a pacemaker.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Glucose | Through study completion, up to 1 year.
  The investigators will measure glucose at baseline and 0.5-, 1-, 2-, 3-, and 4-hours after each meal trial.
Insulin | Through study completion, up to 1 year.
  The investigators will measure serum insulin at baseline and 0.5-, 1-, 2-, 3-, and 4-hours after each meal trial.
Triglycerides | Through study completion, up to 1 year.
  The investigators will measure triglycerides at baseline and 0.5-, 1-, 2-, 3-, and 4-hours after each meal trial.
HDL-C | Through study completion, up to 1 year.
  The investigators will measure HDL-C at baseline and 0.5-, 1-, 2-, 3-, and 4-hours after each meal trial.
Lipopolysaccharide binding protein (LBP) | Through study completion, up to 1 year.
  The investigators will measure serum LBP at baseline and 0.5-, 1-, 2-, 3-, and 4-hours. after each meal trial.
soluble CD14 (sCD14) | Through study completion, up to 1 year.
  The investigators will measure serum sCD14 at baseline and 0.5-, 1-, 2-, 3-, and 4-hours after each meal trial.
Interleukin (IL)-6 | Through study completion, up to 1 year.
  The investigators will measure serum IL-6 at baseline and 0.5-, 1-, 2-, 3-, and 4-hours after each meal trial.
Flow-mediated dilation | Through study completion, up to 1 year.
  The investigators will measure FMD at baseline, 2-hours, and 4-hours after each meal trial.

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Keirns, Principal Investigator — Ball State University
Locations (1):
- Health Professions Building, Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No